CLINICAL TRIAL: NCT01086605
Title: Randomized Phase II Study of Two Doses of Pixantrone in Patients With Metastatic Breast Cancer
Brief Title: Pixantrone Dimaleate in Treating Patients With HER2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N1031; NCCTG-N1031; CDR0000667253 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02021 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: HER2-negative breast cancer; male breast cancer; recurrent breast cancer; stage IV breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive pixantrone dimaleate IV over 1 hour on day 1. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pixantrone dimaleate
- Arm II (Experimental): Patients receive pixantrone dimaleate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pixantrone dimaleate

INTERVENTIONS:
Drug: pixantrone dimaleate — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pixantrone dimaleate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pixantrone dimaleate in different ways may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well pixantrone dimaleate works in treating patients with HER2-negative metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the proportion of confirmed tumor responses at each dose level of pixantrone

Secondary

* To describe the distribution of progression-free survival (PFS) times of patients receiving pixantrone
* To assess the 6-month PFS rate in patients receiving each dose level of pixantrone
* To describe the overall survival distribution of patients receiving pixantrone
* To assess the adverse event profile of pixantrone in the treatment of patients with metastatic breast cancer.
* To evaluate the quality of life and patient-reported symptoms of patients receiving the study regimen

OUTLINE: This is a multicenter study. Patients are randomized according to prior doxorubicin treatment ( yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive pixantrone dimaleate IV over 1 hour on day 1. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive pixantrone dimaleate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Some patients undergo blood sample collection at baseline and periodically during study for circulating tumor cells analysis by CellSearch System and mRNA isolation assays.

Patients complete quality-of-life questionnaires using the Linear Analogue Self Assessment (LASA6) and the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) at baseline and periodically during study.

After completion of study therapy, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
Registration and Randomization - Inclusion Criteria

1. Women or men
2. ≥18 years of age
3. Histologically or cytologically confirmed adenocarcinoma of the breast and clinical evidence of metastatic breast cancer.
4. Pre-treatment requirements:

   4.1. Must have been previously treated in neoadjuvant, adjuvant or metastatic setting with anthracycline and/or taxane.

   4.2. Must have received 2-3 prior chemotherapy treatment regimens NOTE: If NO prior (neo)adjuvant chemotherapy, patient must have received a minimum of 2 prior chemotherapy regimens in the metastatic setting.

   4.2.1 NOTE: If prior (neo)adjuvant chemotherapy HAS been given, patient must have received at least 1 prior chemotherapy regimen in the metastatic setting.

   4.3. Prior hormonal therapy allowed in the neo-adjuvant, adjuvant, or metastatic setting.

   Unlimited prior hormonal therapy is allowed.
5. Patients must have measurable disease as defined in the protocol.
6. Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
7. The following laboratory values obtained ≤15 days prior to registration.

   7.1 Hemoglobin ≥10.0g/dL

   7.2 ANC ≥1500/mm^3

   7.3 Platelet count ≥100,000/mL

   7.4 Total bilirubin ≤1.5 x ULN)

   7.5 SGOT (AST) and SGPT (ALT) ≤5 x ULN

   7.6 Serum creatinine ≤1.5 x ULN
8. LVEF ≥50% and EKG within institutional normal limits completed ≤22 days prior to registration.
9. ECOG Performance Status (PS) of 0, 1 or 2.
10. Life expectancy >3 months
11. Ability to complete questionnaire(s) by themselves or with assistance.
12. Patient has provided written informed consent
13. Willingness to return to NCCTG enrolling institution for follow-up.

Registration and Randomization - Exclusion Criteria

1. Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.

   1.1 Pregnant women

   1.2 Nursing women

   1.3 Men or women of childbearing potential who are unwilling to employ adequate contraception (as determined by the treating physician)
2. Stage III or IV invasive cancer (other than breast cancer) in ≤3 years prior to registration (with the exception of non-melanoma skin cancer).
3. HER2 positive breast cancer (3+ by IHC or FISH amplified) breast cancer by ASCO/CAP guidelines
4. Has already received lifetime cumulative treatment with doxorubicin equivalent to >400 mg/m2.
5. >3 prior chemotherapy regimens for breast cancer.

   5.1 NOTE: This number includes (neo)adjuvant chemotherapy, if given. If (neo)adjuvant chemotherapy HAS been given it counts as one (1) regimen.
6. Major surgery, chemotherapy, or immunologic therapy ≤3 weeks prior to registration.

   6.1 NOTE: If patient has received prior treatment with bevacizumab, treatment on this trial should not begin until ≥4 weeks after the last dose of bevacizumab.
7. Radiotherapy ≤4 weeks prior to registration, except if to a non-target lesion only.

   7.1 Prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.

   7.2 If patient receives single dose radiation for palliation or radiation to non-target lesion, they may immediately proceed to registration without waiting.

   7.3 Acute adverse events from radiation must have resolved to ≤Grade 1 (according to current version of NCI CTCAE).
8. Evidence of active brain metastasis including leptomeningeal involvement.

   8.1 CNS metastasis controlled by prior surgery and/or radiotherapy is allowed. To be considered controlled, there must be at least 2 months of no symptoms or evidence of progression prior to study entry and corticosteroid therapy given to control brain edema must have been discontinued.
9. Uncontrolled hypertension (blood pressure [BP] >160/90mmHg on ≥2 occasions at least 5 minutes apart). (Patients who have recently started or adjusted anti-hypertensive medications are eligible providing that BP is <140/90mmHg on any new regimen for ≥3 different observations in ≥14 days.).
10. Clinically significant cardiovascular or cerebrovascular disease, including any history of the following at any time prior to registration:

    10.1 Myocardial infarction

    10.2 Unstable angina pectoris

    10.3 New York Heart Association (NYHA) Class II or greater congestive heart failure

    10.4. Uncontrolled or clinically significant cardiac arrhythmia (patients with controlled atrial fibrillation are eligible)
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
12. Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
13. History of allergy or hypersensitivity to drug product excipients or agents chemically similar to pixantrone.
14. Currently receiving treatment in a different clinical study in which investigational procedures are performed or investigational therapies are administered.

14.1 Patient may not enroll in such clinical trials while participating in this study.

Exception may be granted for trials related to symptom management (Cancer Control) which do not employ hormonal treatments or treatments that may block the path of the targeted agents used in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2014-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Moreno-Asptia, MD, Study Chair — Mayo Clinic
Locations (230):
- United States (230):
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Comprehensive Cancer Care, PC, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Rutherford Hospital, Rutherfordton, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Willamette Falls Hospital, Oregon City, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Sideras K, Hillman DW, Giridhar K, Ginos BF, Tenglin RC, Liu H, Chen B, Tan W, Gross GG, Mowat RB, Dueck AC, Perez EA, Moreno-Aspitia A. Randomized Phase II Study of Two Doses of Pixantrone in Patients with Metastatic Breast Cancer (NCCTG N1031, Alliance). Oncologist. 2022 Apr 21;27(5):338-e368. doi: 10.1093/oncolo/oyab065. Online ahead of print. PMID 35445723

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I/Group A (Pixantrone IV Day 1): Patients receive 180 mg/m^2 pixantrone dimaleate IV over 1 hour on day 1. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
- Arm II/Group B (Pixantrone IV Days 1, 8, and 15): Patients receive 85 mg/m^2 pixantrone dimaleate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I/Group A (Pixantrone IV Day 1) | Arm II/Group B (Pixantrone IV Days 1, 8, and 15)
Started | 24 | 22
Completed | 24 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I/Group A (Pixantrone IV Day 1) | Arm II/Group B (Pixantrone IV Days 1, 8, and 15) | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Median (Full Range); unit: years] | 56.5 [42 to 79] | 52.5 [38 to 75] | 55.5 [38 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Confirmed Tumor Responses (Complete or Partial Response)
Description: The proportion of confirmed responses will be estimated by the number of women who achieve a CR or PR on two consecutive evaluations at least 6-8 weeks apart depending on the dose level. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients at each dose level. Confidence intervals for the true success proportion at each dose level will be calculated according to the approach of Duffy and Santner. Response will be evaluated in this study using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1); Complete Response (CR): Disappearance of all non-nodal target lesions, each target lymph node must have reduction in short axis to <1.0 cm. and normalization of tumor biomarkers. Partial Response (PR): At least a 30% decrease in the sum of the longest diameters of the non-nodal target lesions and the short axis of the target lymph nodes taking as reference the Baseline Sum of Diameters.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Arm I/Group A (Pixantrone IV Day 1) | Arm II/Group B (Pixantrone IV Days 1, 8, and 15)
Number analyzed (Participants) | 24 | 22
proportion | 0.08 [0.01 to 0.27] | 0.05 [0 to 0.24]

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression the patient will be considered to have had disease progression at the time of their death. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. In the case of a patient starting treatment and then never returning for any evaluations, the patient will be censored for progression one day post-registration. The distribution of time to progression will be estimated using the method of Kaplan-Meier at each dose level. Progression is defined using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1).
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I/Group A (Pixantrone IV Day 1) | Arm II/Group B (Pixantrone IV Days 1, 8, and 15)
Number analyzed (Participants) | 24 | 22
months | 2.8 [1.4 to 7.9] | 2.5 [1.7 to 4.1]

3. Secondary Outcome: 6-month Progression-free Survival Rate
Description: The 6-month progression free survival (6-mo PFS) rate is the proportion of efficacy-evaluable patients progression-free 6 months from registration. The 6-mo PFS rate is defined as the total number of efficacy-evaluable patients on study without documentation of disease progression 6 months from registration divided by the total number of efficacy-evaluable patients enrolled on study. Patients who died without documentation of progression will be considered to have progressed on the date of their death. The true 6-mo PFS rate will be estimated by the proportion of efficacy-evaluable patients on study without documentation of disease progression 6 months from registration at each dose level. Binomial confidence intervals for 6-mo PFS rate will be constructed for each dose level. Progression is defined using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1).
Time Frame: At 6 months
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Arm I/Group A (Pixantrone IV Day 1) | Arm II/Group B (Pixantrone IV Days 1, 8, and 15)
Number analyzed (Participants) | 24 | 22
proportion | 0.375 [0.224 to 0.629] | 0.265 [0.227 to 0.553]

4. Secondary Outcome: Overall Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier at each dose level.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I/Group A (Pixantrone IV Day 1) | Arm II/Group B (Pixantrone IV Days 1, 8, and 15)
Number analyzed (Participants) | 24 | 22
months | 16.8 [9 to NA] — The study did not have enough deaths or patients were not followed long enough to get the upper limit of the 95% confidence interval of median overall survival. | 9.6 [4.7 to NA] — The study did not have enough deaths or patients were not followed long enough to get the upper limit of the 95% confidence interval of median overall survival.

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients with measurable disease who have achieved a confirmed response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented at each dose level. If a patient dies subsequent to the confirmed response without a documentation of disease progression, the patient will be considered to have had disease progression at the time of their death. In the case of a patient failing to return for evaluations before a documentation of disease progression, the patient will be censored for progression on the date of last evaluation. The distribution of duration of response will be estimated using the method of Kaplan-Meier at each dose level.
Time Frame: Up to 5 years
Measure: Mean (Full Range); unit: months
Groups:
- Arm I/Group A + Arm II/Group B: Arm I/Group A: Patients receive 180 mg/m^2 pixantrone dimaleate IV over 1 hour on day 1. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Arm II/Group B: Patients receive 85 mg/m^2 pixantrone dimaleate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I/Group A + Arm II/Group B
Number analyzed (Participants) | 46
months | 5.8 [4.6 to 7.2]

6. Secondary Outcome: Toxicity
Description: For this secondary endpoint, toxicity is defined as a grade 3 or higher adverse events that is classified as either possibly, probably, or definitely related to study treatment. The assignment of attribution to study treatment and grade (or degree of severity) of the adverse event are classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The number of participants reporting a grade 3 or higher toxicity is reported. For a list of all reported adverse events, please refer to the Adverse Events Section below.
Time Frame: Up to 1 year after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I/Group A (Pixantrone IV Day 1) | Arm II/Group B (Pixantrone IV Days 1, 8, and 15)
Number analyzed (Participants) | 24 | 21
Participants | 16 | 19

ADVERSE EVENTS:
Time Frame: Adverse events are assessed within 15 days prior to registration and during the Active Monitoring Phase: less than or equal to 3 days prior to each subsequent cycle of treatment, at end of treatment, and during observation after end of treatment (every 3 months for 1 year).
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All graded adverse events are reported.
Groups:
- Arm I/Group A: Patients receive 180 mg/m^2 pixantrone dimaleate IV over 1 hour on day 1. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
- Arm II/Group B: Patients receive 85 mg/m^2 pixantrone dimaleate IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I/Group A | Arm II/Group B
Serious Adverse Events (participants affected / at risk) | 3/24 | 9/22
Other Adverse Events (participants affected / at risk) | 23/24 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I/Group A (N=24) | Arm II/Group B (N=22)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (3)
White blood cell decreased (Investigations) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I/Group A (N=24) | Arm II/Group B (N=22)
Anemia (Blood and lymphatic system disorders) | 18 (62) | 18 (43)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 2 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (7) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 10 (17) | 6 (7)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 8 (17) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (54) | 16 (25)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 9 (12) | 9 (12)
Chills (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 21 (76) | 20 (49)
Fever (General disorders) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (4)
Malaise (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (6) | 6 (8)
Alkaline phosphatase increased (Investigations) | 1 (1) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 5 (10) | 8 (14)
Blood bilirubin increased (Investigations) | 2 (2) | 4 (4)
Creatinine increased (Investigations) | 2 (9) | 2 (3)
Ejection fraction decreased (Investigations) | 3 (3) | 1 (3)
Lymphocyte count decreased (Investigations) | 2 (5) | 4 (5)
Neutrophil count decreased (Investigations) | 20 (40) | 21 (54)
Platelet count decreased (Investigations) | 5 (10) | 8 (10)
Weight loss (Investigations) | 0 (0) | 2 (5)
White blood cell decreased (Investigations) | 8 (18) | 7 (16)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 3 (10)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 4 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (5)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 5 (10)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (6)
Urine discoloration (Renal and urinary disorders) | 2 (2) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (69) | 16 (41)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 12 (30) | 8 (25)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes